CLINICAL TRIAL: NCT01563887
Title: Identifying Driving Risk Factors in T1DM and Their Reduction Via Behavioral Intervention
Brief Title: Identifying Driving Risk Factors in Type 1 Diabetes and Their Reduction Via Internet Program (DiabetesDriving.Com)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Daniel Cox, PhD, Professor, Department of Psychiatry and NB Sciences, University of Virginia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 15360; 5R01DK028288-25 (NIH)
Record Dates: First submitted 2012-02-29; First posted 2012-03-27 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: Type 1 Diabetes; Hypoglycemia; Driving; Driving safety; Internet; Web; Treatment; Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DD.com (Experimental): Participants in this arm will receive the DiabetesDriving.com internet intervention intended to help reduce their risk of being in a future collision.
  Interventions: Behavioral: DD.com
- DD.com + MI (Experimental): Participants will receive the DiabetesDriving Internet intervention and two 60 minute Motivational Interview (MI) sessions over the telephone. The MI sessions will take place once before and once following completion of the Internet intervention. This interview will focus on making explicit individual's ambivalence around changing behavior.
  Interventions: Behavioral: DD.com + MI

INTERVENTIONS:
Behavioral: DD.com — Internet intervention in which participants will complete 6 Cores, or classes over the internet, focusing on risk factors and prevention, detection, and management of hypoglycemia before and while driving.
  Arms: DD.com
Behavioral: DD.com + MI — Prior to starting and immediately after finishing the DiabetesDriving.com internet intervention, a one hour motivational interview will be conducted with participants. Internet intervention in which participants will complete 6 Cores, or classes over the internet, focusing on risk factors and prevention, detection, and management of hypoglycemia before and while driving.
  Arms: DD.com + MI

SUMMARY:
This study will recruit drivers with Type 1 diabetes from across the U.S. and assign them to four groups based on their presumed risk level- routine care low risk, routine care high risk, or to one of two Internet interventions focused on reducing hypoglycemia driving. All subjects will be followed for two years to determine whether and which intervention was most effective at reducing hypoglycemia related driving collisions.

DETAILED DESCRIPTION:
The investigators have demonstrated that drivers with Type 1 diabetes have at least twice as many collisions as their non-diabetic spouses, that about half of drivers with Type 1 diabetes have at least one hypoglycemic driving mishap a year, and 5% have at least six such events in a year. However, at this point the investigators can not accurately predict those individuals who will have hypoglycemia driving mishaps, which is one goal of this study. The investigators have also demonstrated that face-to-face behavioral interventions focusing on reducing the occurrence of hypoglycemia have lead to significantly fewer vehicular collisions and citations. The question arises whether such a behavioral intervention, specifically focused on reducing hypoglycemia while driving, can be effectively delivered over the internet.

Participants will first complete an Interest form. This questionnaire is used to determine an individual's presumed risk category (high or low risk). Research staff will use the risk category to randomly assign participants to one of four groups according to the randomization scheme. The four groups include: 1) Routine Care - low risk, 2) Routine Care - high risk, 3) DiabetesDriving.com (DD.com) where they will participate in an Internet intervention, 4) DiabetesDriving.com + Motivational Interviewing (MI) where subjects will receive the Internet intervention and two 60 minute MI sessions over the telephone. The MI sessions will take place once before and once following completion of the Internet intervention (within 7 days). This interview will focus on making explicit individuals' ambivalence around changing behavior.

Individuals assigned to the DD.com and DD.com+MI groups will complete 6 Cores, or classes over the internet, focusing on risk factors and prevention, detection, and management of hypoglycemia before and while driving. Each core will take approximately 30 minutes to complete. Core 0 is a tutorial on how to use the internet program. Core 1 focuses on how to use the Tool Kit; Core 2 focuses on how to be a safer driver in general; Core 3 focuses on how to prevent hypoglycemia from occurring while driving; Core 4 focuses on detecting and treating hypoglycemia during a drive; Core 5 focuses on how to maintain the improvements they have achieved in the previous Core over the next 12 months.

After completing a Core, individuals must wait a week before they can start the next Core. During this time individuals will complete at least three Daily Progress Notes, where they will rate their success at achieving their driving goals established in the previous Core. The Cores will take up to 8 weeks to complete before completing Driving Survey 2.

All participants will complete Driving Surveys and monthly driving diaries. The first Driving Survey (Driving Survey 0) will be available to participants as soon as they are consented. Driving Surveys will then be given at 2 and 14 months after submission of Driving Survey 0. Participants will also complete monthly driving diaries, where they will report their driving experiences for the full previous month. Monthly driving diaries will be available on the first day of the next full month 98 days (14 weeks) after completing the Driving Survey at month 2 and continue for 12 months. Twenty-six months after submitting Driving Survey 0, participants will be emailed for a two year follow-up. They will be asked to complete a brief questionnaire on driving outcomes (collisions, citations, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Have been diagnosed with Type 1 diabetes for at least one year
2. Started taking insulin less than a year after being diagnosed with Type 1 diabetes
3. Measure blood glucose at least twice a day
4. Legal and valid driver's license
5. Drives greater than 5,000 per year
6. Regular access to the Internet, either through family computer or another readily accessible computer
7. Age 18 - 70 years
8. English speaker

Exclusion Criteria:

1. Type 2 diabetes
2. Does not take insulin
3. Does not drive
4. Does not have legal and valid driver's license
5. Does not have routine access to the internet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The change in the number of hypoglycemia-related driving mishaps | 10 weeks and 62 weeks after submitting the first Driving Survey
  Driving Surveys will be completed prior to study initiation, immediately after the intervention is finished, and again in one year. Monthly Driving Diaries will be completed each month for the year after the intervention finishes beginning 14 weeks after submitting the first Driving Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cox, Ph.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Cox DJ, Gonder-Frederick LA, Singh H, Ingersoll KS, Banton T, Grabman JH, Schmidt K, Clarke W. Predicting and Reducing Driving Mishaps Among Drivers With Type 1 Diabetes. Diabetes Care. 2017 Jun;40(6):742-750. doi: 10.2337/dc16-0995. Epub 2017 Apr 12. PMID 28404657